CLINICAL TRIAL: NCT01863316
Title: The Comparison of the Clinical Efficacy Between I-gel and LMA-Supreme, the Two Most Recently Developed Supraglottic Airway Devices, in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1-2013-0023
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Elective Surgery of Short Duration (Less Than 2 hr) Undergoing General Anesthesia Using Supraglottic Airway
Keywords: LMA Supreme, i-gel, supraglottic airway

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1) I gel group (Experimental): using supraglottic airway I gel
  Interventions: Device: I gel
- 2) LMA Supreme group (Active Comparator): using supraglottic airway LMA Supreme
  Interventions: Device: LMA Supreme

INTERVENTIONS:
Device: I gel
  Arms: 1) I gel group
Device: LMA Supreme
  Arms: 2) LMA Supreme group

SUMMARY:
Although the safety and efficacy of the I gel in children has been shown in several large observational studies, There is no study about comparison of the clinical efficacy between I-gel and LMA-Supreme , in particular sizes 1 and 1½. The pediatric i-gel and LMA Supreme are new supraglottic airway device for children. It is made of a soft, gel-like elastomer with a noninflatable cuff. Studies about I-gel and LMA Supreme in adults have been promising, showing an easy insertion, high airway leak pressures, and low complication rates with few postoperative complaints. The aim of this study is to compare clinical performance of the pediatric i-gel and LMA Supreme in infants.

ELIGIBILITY:
Inclusion Criteria:

1. Infants (0-1 year of age) scheduled for elective surgery of short duration (less than 2 hr) undergoing general anesthesia using supraglottic airway

Exclusion Criteria:

1. Patients with an abnormal airway, reactive airway disease, gastroesophageal reflux disease, chronic respiratory disease, or a history of an upper respiratory tract infection in the preceding 6-week period

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
airway leak pressure | within 5 min of insertion of each device
  Airway leak pressure was determined by adjusting the expiratory valve of the breathing circle to 30 cmH2O (fixed fresh gas flow 3 L/min) and recording the pressure when equilibrium was reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei University College of Medicine, Seoul, Seoul, South Korea